CLINICAL TRIAL: NCT00052286
Title: A Pilot Study of Modafinil for Treatment of Fatigue and Neurobehavioral Dysfunction in Adult Brain Tumor Patients
Brief Title: Modafinil in Treating Fatigue and Behavioral Change in Patients With Primary Brain Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000258139; UCLA-0206017; CEPHALON-UCLA-0206017; NCI-G02-2133
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2016-02

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Fatigue
Keywords: adult brain tumor; fatigue; cognitive/functional effects
MeSH Terms: conditions — Central Nervous System Neoplasms; Fatigue; Brain Neoplasms | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug dosage 1 (Experimental): - Arm I: Patients receive oral high-dose modafinil twice daily.
  Interventions: Drug: modafinil
- drug dosage 2 (Experimental): - Arm II: Patients receive oral low-dose modafinil twice daily.
  Interventions: Drug: modafinil

INTERVENTIONS:
Drug: modafinil

SUMMARY:
RATIONALE: Modafinil may be effective in relieving fatigue and improving behavioral changes such as memory loss in patients who have undergone treatment for primary brain cancer. The effectiveness of modafinil in relieving fatigue and improving behavioral change is not yet known.

PURPOSE: This randomized clinical trial is comparing how well two different doses of modafinil work in treating fatigue and behavioral changes in patients who have undergone treatment for primary brain cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of low-dose vs high-dose modafinil for treatment of fatigue and neurobehavioral dysfunction in patients with primary brain tumors.
* Determine the safety of this drug in these patients.
* Compare quality of life of patients treated with 2 different doses of this drug.

OUTLINE: This is a randomized, double-blind, parallel-group study. Patients are randomized to 1 of 2 arms.

* Randomized phase:

  * Arm I: Patients receive oral high-dose modafinil twice daily.
  * Arm II: Patients receive oral low-dose modafinil twice daily. In both arms, treatment in this phase continues for 3 weeks followed by a 1-week washout period.
* Extended treatment phase:After the 1-week washout period, all patients receive oral low-dose modafinil once daily on days 1-3. The dose is then titrated to an optimal level and administered in divided doses.

Fatigue, neurobehavioral dysfunction, and quality of life are assessed during the randomized phase at baseline and on days 7 and 21 and then during the extended treatment phase at baseline and on days 28 and 56.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary malignant brain tumor and receiving treatment in the UCLA Neuro-Oncology Program
* Nonmalignant cerebral tumors also allowed
* Received some combination of prior therapy for disease, including neurosurgical resection, radiotherapy, and cytotoxic or cytostatic chemotherapy
* Mild to severe fatigue and/or attention/memory impairment, as measured by the Clinical Global Impression of Severity Scale
* Age 21 to 65
* Able to speak English
* Capable of completing self-rating scales and one-on-one psychometric tests
* Negative pregnancy test
* Fertile patients must use effective contraception
* Concurrent conventional chemotherapy (e.g., carboplatin, lomustine, temozolomide) allowed
* Concurrent glucocorticoids (e.g., dexamethasone) allowed
* Concurrent tamoxifen allowed
* At least 30 days since prior stimulants (e.g., amphetamines or methylphenidate)
* Concurrent anticonvulsants allowed
* Concurrent isotretinoin allowed

Exclusion Criteria:

* Have significant hepatic disease, defined as SGOT greater than or equal to 2.5 times the upper limit of normal.
* Have significant renal disease, defined as creatinine greater than or equal to 1.5mg/dl.
* severe cognitive impairment
* other terminal illness
* emergency patient
* institutional resident
* prisoner or parolee
* UCLA students or staff
* pregnant or nursing
* concurrent irinotecan
* concurrent participation in UCLA experimental chemotherapy trials
* prior modafinil
* concurrent experimental anticancer medication
* concurrent tricyclic antidepressants and/or monoamine oxidase inhibitors

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-09; Primary Completion 2006-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Neurocognitive functioning | at baseline and weeks 1, 3, 4, 8, and 10

SECONDARY OUTCOMES:
Global functioning as assessed by Clinical Global Impression of Severity and Clinical Global Impression of Change. | at baseline and weeks 1, 3, 4, 5, 7, 8, 9, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Cloughesy, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States